CLINICAL TRIAL: NCT02536638
Title: Quantitating Proteinuria During Acute Pyelonephritis In Pregnancy
Brief Title: Proteinuria During Acute Pyelonephritis In Pregnancy
Status: Completed | Type: Observational
Sponsor: MemorialCare Health System (Other)
Responsible Party: Principal Investigator, Kenneth Chan, MD, Maternal Fetal Medicine, MemorialCare Health System
Other Study IDs: 510-15
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Proteinuria
Keywords: urine protein; pregnancy; pyelonephritis; kidney infection
MeSH Terms: conditions — Proteinuria; Pyelonephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine collection for 24 hour urine protein and creatinine analysis urine sample for urinalysis with microscopy and culture blood for measurement of serum creatinine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pyelonephritis Group: patients with pyelonephritis
  Interventions: Other: Exposure to pyelonephritis
- Without pyelonephritis Group: patients without pyelonephritis

INTERVENTIONS:
Other: Exposure to pyelonephritis — Pyelonephritis group are patients with exposure to pyelonephritis Without pyelonephritis group are patients without pyelonephritis
  Groups: Pyelonephritis Group

SUMMARY:
The purpose of this research study is to compare the amount of protein excreted by the kidneys in a 24-hour period between patients who have a kidney infection and those who do not have a kidney infection.

DETAILED DESCRIPTION:
Preeclampsia is a pregnancy-unique disorder that is cured only with delivery of the baby, even if the pregnancy is premature. Defined by both blood pressure and proteinuria criteria, diagnosis is often obscured by renal processes like systemic lupus erythematosus or nephrotic syndrome that increase urinary protein spillage. Proteinuria is defined as a total protein urinary excretion exceeding 300 mg in a 24-hour urine collection in pregnancy. This is suggested to be double the protein excretion in the non-pregnancy population at 150 mg/day. A mean 24-hour urine protein excretion of 204.3 mg (± 92.5) was found in the non-hypertensive pregnant population.

Physiological changes in pregnancy predispose patients to urinary tract infections; ureteral compression by the gravid uterus, progesterone-mediated slowing of ureteral peristalsis and decreased bladder tone, and mechanical compression of the bladder contribute to impaired clearance of bacteria from the urinary tract. Indeed, acute cystitis complicates 2-4% of all pregnancies. While it has been said that urinary tract infections increase proteinuria, it is unknown how much protein spillage should be expected in the general or the pregnant populations. Hence a patient with pyelonephritis may obscure the diagnosis of preeclampsia if she spills urinary protein from her infection.

The purpose of this study is to compare the mean of 24-hour urine protein in pregnant patients with and without acute pyelonephritis.

The importance of this study will be to determine if urine protein excretion is in fact increased in the setting of pyelonephritis. This will allow for reliable evaluation of urine protein during the work up for preeclampsia in those women also found having a kidney infection.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old admitted at Miller Children and Women's Hospital Long Beach Memorial Medical Center
* Gestational age between 20 weeks and 0 days to 41 weeks and 0 days
* Singleton pregnancy
* Pyelonephritis group:

meeting 2 out of 3 criteria:

1. Fever > 100.4
2. Costovertebral angle tenderness
3. Positive urine culture - without pyelonephritis group: without acute cystitis and pyelonephritis

Positive culture defined as: quantitative count of ≥ 100,000 CFU/mL or single catheterized urine specimen with quantitative count of 100 CFU/mL.

Exclusion Criteria:

* Chronic hypertension
* Pre-gestational diabetes
* Autoimmune disorders
* Preexisting renal disease
* Multiple gestation
* Vaginal bleeding
* Preeclampsia
* Hospital admission > 3 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to inpatient management of acute pyelonephritis meeting the inclusion and exclusion criteria will be enrolled in the study. A 24 hour urine collection with be performed for evaluation of protein.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
24-hour urine protein | 7 days
  urine protein will be measured upon patient enrollment to the study (i.e. during the study enrollment hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chan, MD, Principal Investigator — Maternal Fetal Medicine
Locations (1):
- Miller Children's and Women's Hospital at Long Beach Memorial Medical Center, Long Beach, California, United States

REFERENCES:
- [Background] Lindheimer MD, Kanter D. Interpreting abnormal proteinuria in pregnancy: the need for a more pathophysiological approach. Obstet Gynecol. 2010 Feb;115(2 Pt 1):365-375. doi: 10.1097/AOG.0b013e3181cb9644. PMID 20093912
- [Background] Osmundson SS, Lafayette RA, Bowen RA, Roque VC, Garabedian MJ, Aziz N. Maternal proteinuria in twin compared with singleton pregnancies. Obstet Gynecol. 2014 Aug;124(2 Pt 1):332-337. doi: 10.1097/AOG.0000000000000383. PMID 25004349
- [Background] Gilstrap LC 3rd, Ramin SM. Urinary tract infections during pregnancy. Obstet Gynecol Clin North Am. 2001 Sep;28(3):581-91. doi: 10.1016/s0889-8545(05)70219-9. PMID 11512502
- [Background] Jolley JA, Wing DA. Pyelonephritis in pregnancy: an update on treatment options for optimal outcomes. Drugs. 2010 Sep 10;70(13):1643-55. doi: 10.2165/11538050-000000000-00000. PMID 20731473
- [Background] Carter JL, Tomson CR, Stevens PE, Lamb EJ. Does urinary tract infection cause proteinuria or microalbuminuria? A systematic review. Nephrol Dial Transplant. 2006 Nov;21(11):3031-7. doi: 10.1093/ndt/gfl373. Epub 2006 Jul 22. No abstract available. PMID 16861738
- [Background] Rubin RH, Shapiro ED, Andriole VT, Davis RJ, Stamm WE. Evaluation of new anti-infective drugs for the treatment of urinary tract infection. Infectious Diseases Society of America and the Food and Drug Administration. Clin Infect Dis. 1992 Nov;15 Suppl 1:S216-27. doi: 10.1093/clind/15.supplement_1.s216. PMID 1477233
- [Background] Nicolle LE, Bradley S, Colgan R, Rice JC, Schaeffer A, Hooton TM; Infectious Diseases Society of America; American Society of Nephrology; American Geriatric Society. Infectious Diseases Society of America guidelines for the diagnosis and treatment of asymptomatic bacteriuria in adults. Clin Infect Dis. 2005 Mar 1;40(5):643-54. doi: 10.1086/427507. Epub 2005 Feb 4. No abstract available. PMID 15714408
- [Background] CLARK LC, THOMPSON H, BECK EI. The excretion of creatine and creatinine during pregnancy. Am J Obstet Gynecol. 1951 Sep;62(3):576-83. doi: 10.1016/0002-9378(51)91156-8. No abstract available. PMID 14877920
- [Result] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027